CLINICAL TRIAL: NCT00577200
Title: The Safety of Driving in Patients After Minor Surgery With Monitored Anesthesia Care
Brief Title: Safety of Driving After Minor Surgery With Monitored Anesthesia Care
Acronym: MACDrive
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Asokumar Buvanendran, Principal Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABuv110507
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Minor Surgical Procedures With Monitored Anesthesia Care; Driving Performance After Minor Ambulatory Surgery
MeSH Terms: interventions — Midazolam; Sufentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Control group subjects are not undergoing any surgical procedures and will not be randomized to any anesthetic drug group.
- Midazolam + Sufentanil + Propofol (Experimental): Midazolam 0.03 mg/kg + Sufentanil 0.1 µg/kg + Propofol bolus of 300 µg/kg + infusion at 75 µg/kg/min.
  "For subjects who are chronic pain patients undergoing minor surgical procedures."
  Interventions: Drug: Midazolam; Drug: Sufentanil; Drug: Propofol
- Midazolam and Sufenatnil (Experimental): Midazolam 1-5 mg in holding area + Sufentanil 5-10 mcg.
  "For subjects who are chronic pain patients undergoing minor surgical procedures."
  Interventions: Drug: Midazolam; Drug: Sufentanil

INTERVENTIONS:
Drug: Midazolam — Midazolam
  Other Names: Dormicum, Hypnovel, Midacum, Versed
  Arms: Midazolam + Sufentanil + Propofol; Midazolam and Sufenatnil
Drug: Sufentanil — Sufentanil
  Other Names: Sufenta
  Arms: Midazolam + Sufentanil + Propofol; Midazolam and Sufenatnil
Drug: Propofol — Propofol bolus of 300 µg/kg + infusion at 75 µg/kg/min.
  Other Names: Diprivan
  Arms: Midazolam + Sufentanil + Propofol

SUMMARY:
Patients are currently advised to refrain from driving motor vehicles or using public transportation unescorted for a 24 hour period if they undergo any minor ambulatory surgical procedure with monitored anesthesia care (MAC).However, recently introduced short-acting anesthetics may facilitate rapid recovery and an early return to normal daily activities. The proposed study will compare newer short-acting anesthetic agents (propofol, benzodiazepine, opioid) utilized in MAC, to determine if a particular pharmacological agent, or a combination of agents, impair driving performance as evaluated by driving simulator assessment, at time of discharge from the ambulatory center after minor surgical procedures.Subjects will be grouped as patients with chronic pain undergoing procedures and those without chronic pain undergoing procedures. Subjects with pain issues will be randomized with either 1)Midazolam + Sufentanil + Propofol or 2)Midazolam + Sufentanil. There will be a third group of subjects who are controls not undergoing any procedures.

DETAILED DESCRIPTION:
Patients are currently advised to refrain from driving motor vehicles or using public transportation unescorted for a 24 hour period if they undergo any minor ambulatory surgical procedure with monitored anesthesia care (MAC).However, recently introduced short-acting anesthetics may facilitate rapid recovery and an early return to normal daily activities. The proposed study will compare newer short-acting anesthetic agents (propofol, benzodiazepine, opioid) utilized in MAC, to determine if a particular pharmacological agent, or a combination of agents, impair driving performance as evaluated by driving simulator assessment, at time of discharge from the ambulatory center after minor surgical procedures.The three critical measures of driving performance selected are: weaving, reaction time, and number of collisions. If any of the experimental MAC conditions shows statistical equivalence at discharge with baseline, for all three criterion measures, then that anesthetic regimen can be designated as "safe to drive". If this study can demonstrate such an early recovery of driving ability, which is probably the most complex and dangerous activity commonly encountered, this begs the re-examination of all post-operative activity restrictions imposed on this patient population. Subjects will be grouped as patients with chronic pain undergoing procedures and those without chronic pain undergoing procedures.Subjects with pain issues will be randomized with either 1)Midazolam + Sufentanil + Propofol or 2)Midazolam + Sufentanil. There will be a third group of subjects who are controls not undergoing any procedures.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory surgical patient possessing a valid driving license and presenting for a minor procedure that does not physically impact ability to drive (such as hand, arm, and lower extremity surgery).
* Another group of subjects who are not scheduled for a procedure will be given a driving simulator exercise and they will be control group.

Exclusion Criteria:

* Any surgical case that lasted more than one hour and required general anesthesia will be excluded.
* Patients with a history of chronic benzodiazepine or alcohol abuse, alcohol or other substance dependence or recent use of medications with sleep altering qualities, and driving simulator sickness.
* Patients who cannot follow a simple driving task and cannot sit on a chair for the driving test due to medical conditions will also be excluded.
* History of seizures

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 625 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Weaving, measured as the standard deviation of lateral position. | 6 h

SECONDARY OUTCOMES:
Reaction time (RT) | 6 h

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, M.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States